CLINICAL TRIAL: NCT02729766
Title: Effects of Empagliflozin an SGLT2-Inhibitor on Healthy Volunteers With Induced Hypotonic Hyponatremia - the DIVE Study
Acronym: DIVE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-00024
Record Dates: First submitted 2016-03-24; First posted 2016-04-06 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Inappropriate ADH Syndrome
Keywords: Hyponatremia; SGLT2 inhibitor
MeSH Terms: conditions — Inappropriate ADH Syndrome; Hyponatremia | interventions — empagliflozin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Empagliflozin 25mg Tbl (Active Comparator): Induced hypotonic hyponatremia - SIAD model: Hypotonic hyponatremia will be induced in healthy volunteers through oral overhydration and parenteral administration of desmopressin (Minirin)® 4ug. After administration of the study drug, the artificial SIAD will be sustained with infusion of hypotonic sodium-solution (NaCl 0.45%) over two hours.
  Interventions: Other: Induced hypotonic hyponatremia - SIAD model; Drug: Empagliflozin 25mg Tbl
- Placebo P-Tablet (Placebo Comparator): Induced hypotonic hyponatremia - SIAD model: Hypotonic hyponatremia will be induced in healthy volunteers through oral overhydration and parenteral administration of desmopressin (Minirin)® 4ug. After administration of the study drug, the artificial SIAD will be sustained with infusion of hypotonic sodium-solution (NaCl 0.45%) over two hours.
  Interventions: Other: Induced hypotonic hyponatremia - SIAD model; Drug: Placebo P-Tablet

INTERVENTIONS:
Other: Induced hypotonic hyponatremia - SIAD model
  Other Names: Induced hypotonic hyponatremia
Drug: Empagliflozin 25mg Tbl
  Arms: Empagliflozin 25mg Tbl
Drug: Placebo P-Tablet
  Arms: Placebo P-Tablet

SUMMARY:
Empagliflozin (Jardiance)® is a sodium glucose co-transporter 2 (SGLT2)-Inhibitor, which is a new treatment option developed for patients with diabetes mellitus type 2. The SGLT2 is expressed in the proximal tubule and reabsorbs approximately 90 percent of the filtered glucose. The inhibition of SGLT2 results in renal excretion of glucose with subsequent osmotic diuresis. This mechanism could result in a therapeutic effect in patients with hypotonic hyponatremia as in the syndrome of inappropriate antidiuretic hormone (ADH) secretion (SIAD). Because patients with SIAD usually have several comorbidities and different medications, studies investigating the physiological effects are difficult to interpret. Therefore a model to study the possible physiological effect of SGLT2-inhibitors in hypotonic hyponatremia as in SIAD is needed.

The aim of this study is to evaluate whether empagliflozin (Jardiance)® has an effect on serum sodium levels of healthy volunteers with induced hypotonic hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Age 18 to 65 years
* serum sodium level 135-145mmol/l
* clinically euvolemic status

Exclusion Criteria:

* Known or suspected allergy to trial product or related products
* Pregnancy or breast feeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* untreated hypothyroidism
* cortisol deficiency
* history of heart failure
* liver cirrhosis at any stage
* kidney disease (GFR <60ml/min)
* epileptic seizures within the last year
* uncontrolled hypertension (systolic blood pressure >160mmHg)
* Diabetes mellitus type 1 or 2
* BMI <18 or >29kg/m2
* other severe disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the area under the curve (AUC) of the serum sodium concentration between time points 2 and 8 hours after administration of the study drug. | concentration measured every hour within 8 hours after drug administration on both study days

SECONDARY OUTCOMES:
Serum sodium concentration at every time point of the study | every hour for twelve hours on each of the two study days
Amount of urinary excretion | every 2 hours for twelve hours on each of the two study days
Serum osmolality at every time point of the study | every hour for twelve hours on each of the two study days
Serum glucose at every time point of the study | every hour for twelve hours on each of the two study days
Urinary osmolality | every two hours for twelve hours on each of the two study days
Urinary glucose | every 2 hours for twelve hours on each of the two study days
Serum electrolytes at time point -1, 0, 2 and 8 | 1 hour before induction of siad, at baseline, 2 hours and 8 hours after administration of study medication on each study day
Urinary electrolytes at time point -1, 0, 2 and 8 | 1 hour before induction of siad, at baseline, 2 hours and 8 hours after administration of study medication on each study day
Plasma level of Copeptin at time point -1, 0, 2 and 8 | 1 hour before induction of siad, at baseline, 2 hours and 8 hours after administration of study medication on each study day
Plasma level of Aldosterone at time point -1, 0, 2 and 8 | 1 hour before induction of siad, at baseline, 2 hours and 8 hours after administration of study medication on each study day
Plasma level of Renin at time point -1, 0, 2 and 8 | 1 hour before induction of siad, at baseline, 2 hours and 8 hours after administration of study medication on each study day
Plasma Level of atrial natriuretic peptide (ANP) at time point -1, 0, 2 and 8 | 1 hour before induction of siad, at baseline, 2 hours and 8 hours after administration of study medication on each study day
Plasma levels of brain natriuretic peptide (BNP) at time point -1, 0, 2 and 8 | 1 hour before induction of siad, at baseline, 2 hours and 8 hours after administration of study medication on each study day
Body weight at every time point of the study | every hour during 12 hours on each of the two study days
Blood pressure at every time point of the study | every hour during 12 hours on each of the two study days
Heart rate at every time point of the study | every hour during 12 hours on each of the two study days
Symptoms of hyponatremia assessed by visual analogue scale (VAS) at every time point of the study | every hour during 12 hours on each of the two study days
Urinary sodium level | every 2 hours for twelve hours on each of the two study days

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof., Principal Investigator — Deputy chief division endocrinology university hospital basel
Locations (1):
- Department Endocrinology University Hospital Basel, Basel, Basel, Switzerland